CLINICAL TRIAL: NCT04962425
Title: Risk Assessment Model of Trastuzumab-related Cardiotoxicity in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Cardiotoxicity study
Record Dates: First submitted 2021-06-27; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-01

CONDITIONS: Cardiac Toxicity; Antitumor Drugs; Breast Cancer
Keywords: Cardiac Toxicity; Antitumor drugs; Breast Cancer; Trastuzumab
MeSH Terms: conditions — Cardiotoxicity; Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The case group: Trastuzumab for the treatment of breast cancer patients with cardiotoxicity.
  Interventions: Drug: Trastuzumab
- The control group: Trastuzumab is used to treat patients with breast cancer who do not present with cardiotoxicity
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab [Herceptin] is a recombinant DNA-humanized monoclonal antibody that selectively targets the HER-2 receptor on the surface of tumor cells.

SUMMARY:
According to the existing clinical data in our hospital, retrospective study was conducted to screen the risk factors with predictive value for TRC(trastuzumab-related cardiotoxicity) risk, and to construct the risk prediction model for TRC.

DETAILED DESCRIPTION:
The breast cancer patients with cardiotoxicity caused by trastuzumab were selected as the case group, and the breast cancer patients without cardiotoxicity were selected as the control group. The clinical baseline data, echocardiographic parameters and serum markers of the case group and the control group were compared to find out the risk factors that may have predictive value for the risk of TRC. The target factors were analyzed by univariate analysis and multivariate Logistic regression analysis, and the TRC risk prediction model was established.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients diagnosed with HER2-positive breast cancer treated in our hospital.
2. Surgical treatment combined with chemotherapy or radiotherapy was completed according to NCCN guidelines, and trastuzumab standard treatment was received for at least half a year.

(3) Cardiac function (including echocardiography or biomarkers) was assessed at least once within 3 months before trastuzumab treatment, and at least once during or after treatment was performed for heart-related tests.

(4) Complete case data.

Exclusion Criteria:

1. Patients who have not been properly treated with trastuzumab or have been treated for less than half a year;
2. Patients who did not receive cardiac function assessment before trastuzumab treatment, during or after treatment;
3. Patients whose case data were missing or lost to follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects were women aged >18 years, diagnosed with HER2-positive breast cancer and already receiving trastuzumab treatment.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac toxicity | 12 months
  The asymptomatic LVEF decreases ≥ 10% of the baseline value or to an absolute value < 50%
Cardiac toxicity | 12 months
  acute or chronic heart failure
Cardiac toxicity | 12 months
  New or aggravated arrhythmias or coronary heart disease
Cardiac toxicity | 12 months
  Myocardial infarction or other cardiac death

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided